CLINICAL TRIAL: NCT02885662
Title: A Study of CS-3150 to Evaluate Efficacy and Safety in Patients With Primary Aldosteronism
Brief Title: Study of CS-3150 in Patients With Primary Aldosteronism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS3150-A-J307
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2017-08

CONDITIONS: Primary Aldosteronism
Keywords: Primary aldosteronism; Hypertension; mineralocorticoid receptor antagonist; Developmental Phase III
MeSH Terms: conditions — Hyperaldosteronism; Hypertension | interventions — esaxerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CS-3150 (Experimental): CS-3150 2.5 to 5.0 mg , orally, once daily after breakfast for 12 weeks.
  Interventions: Drug: CS-3150

INTERVENTIONS:
Drug: CS-3150 — CS-3150 2.5 to 5.0 mg , orally.

SUMMARY:
To examine antihypertensive effect and safety of CS-3150 in patients with primary aldosteronism.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 20 years or older at informed consent
* Patients diagnosed primary aldosteronism by screening test of plasma aldosterone concentration (PAC) and aldosterone to renin ratio (ARR), and confirmatory testing
* Patients satisfying following blood pressure;

  * sitting systolic blood pressure (SBP) ≥ 140 mmHg and <180 mmHg
  * sitting diastolic blood pressure (DBP) ≥ 90 mmHg and <110 mmHg

Exclusion Criteria:

* Secondary hypertension except primary aldosteronism or hypertensive emergency
* Patients diagnosed diabetic nephropathy
* Patients with type 1 diabetes
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2
* Serum potassium level < 3.0 or ≥ 5.1 milliequivalent (mEq)/L

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sitting blood pressure | Baseline to end of Week 12
  Change from baseline in sitting systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Time course of sitting blood pressure | Baseline to end of Week 12
  Time course of sitting systolic and diastolic blood pressure
Proportion of patients achieving sitting blood pressure goal | Baseline to end of Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Japan Organaization of Occupational Health and Safety(JOHAS), Yokohama Rosai Hospital, Yokohama, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/